CLINICAL TRIAL: NCT01061866
Title: Treatment of Refractory Epilepsy With Thalidomide: an Open Trial
Brief Title: Thalidomide Low Threshold in Epilepsy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Neurology and Neurosurgery, Mexico (Other)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Julio Sotelo, MD, National Institute of Neurology and Neurosurgery, Mexico
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INNN 36/06
Record Dates: First submitted 2009-02-17; First posted 2010-02-03 (Estimated); Results first posted 2010-02-03 (Estimated); Last update posted 2010-02-18 (Estimated); Status verified 2009-12

CONDITIONS: Refractory Epilepsy
Keywords: Thalidomide; Antiepileptic drugs; Refractory epilepsy; Sedative drugs
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thalidomide (Experimental): Open-labeled preliminary trial
  Interventions: Drug: 3-phthalimidoglutarimide (Thalidomide)

INTERVENTIONS:
Drug: 3-phthalimidoglutarimide (Thalidomide) — Thalidomide at 200 mg dosage bid was administered during a twelve month period.
  Other Names: Talizer; 3-phthalimidoglutarimide

SUMMARY:
The purpose of this study is to determine whether thalidomide is effective in the refractory epilepsy treatment.

DETAILED DESCRIPTION:
Seven male patients with chronic, refractory epilepsy were included in the present study; in all cases antiepileptic treatment with multiple antiepileptic drugs had been unsuccessful in reducing the frequency or the intensity of seizures. Patients selected for this study were all males due to the high risk of thalidomide for teratogenicity in pregnant women; besides this drawback, thalidomide presents a fair tolerance profile in humans treated with low doses. Informed consent was obtained on each case by the patient and his legal guardian. The protocol was approved by the committees of research and ethics.

Treatment with thalidomide at 200 mg dosage twice daily was administered during a twelve month period. Electroencephalograms were obtained prior and at six months of thalidomide therapy; number and intensity of seizures were individually recorded in a diary by a caregiver (in most cases the patient's mother); signs of neuropathy, a frequent side-effect of chronic thalidomide therapy, were evaluated along the treatment; drowsiness and sedation, which are also common side-effects, were also recorded.

Patients were seen once a week during the treatment period at the Epilepsy Clinic of the National Institute of Neurology and Neurosurgery of Mexico. Once informed consent was obtained, all patients were given seizure diaries to be filled for three months before starting the treatment with thalidomide. Comparisons in the frequency of seizures were made on each patient by contrasting the three months previous to the beginning of thalidomide therapy with the twelve months of the drug trial. One patient (case 6) withdrew from the trial after seven months of thalidomide therapy due to sedation. Another patient (case 7) withdrew from the trial after 3 months of treatment due to exacerbation of seizures as narrated by his mother.

The same schedule of antiepileptic therapy was taken by each patient during three months prior to thalidomide administration and continued it without modification along the trial; therefore, bias due to changes in the associated antiepileptic medications were prevented and each patient served as his own control; so that the effect of thalidomide on the frequency and intensity of seizures could be reasonably evaluated. Thalidomide was purchased by the National Institute of Neurology and Neurosurgery of Mexico at regular price in the pharmaceutical market. No pharmaceutical company participated in any form in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Refractory Epilepsy, males

Exclusion Criteria:

* Females, peripheric neuropathy

Ages: 17 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2006-06; Primary Completion 2007-06 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julio Sotelo, MD, Principal Investigator — National Institute of Neurology and Neurosurgery of Mexico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with refractory epilepsy, 25 years old mean, with antiepileptic treatment and several seizures by month and male gender and they were recruited by Epilepsy Clinic
Pre-assignment Details: Males without seizures three months prior to thalidomide administration and patients without electroencephalographic study and without antiepileptic treatment.
Groups:
- Thalidomide: Thalidomide tablets 200 mg per day during twelve months was administrated to 7 males with 25 years old mean and refractory epilepsy, without modifying their previous treatment.
Period: Overall Study
Arm/Group | Thalidomide
Started | 7
Completed | 5
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Groups:
- Thalidomide: Tablets thalidomide at 200 mg dosage 100 mg in the morning and 100 mg in the night was administered daily during a twelve month period.
Arm/Group | Thalidomide
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 6
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 25 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Mean Number of Daily Seizures at 1 Year.
Time Frame: Baseline 3 months and 1 year of treatment
Population: males of 25 years old mean with refractory epilepsy, antiepileptic treatment and electroencephalographic study
Measure: Mean (Standard Error); unit: Number of Seizures
Arm/Group | Thalidomide
Number analyzed (Participants) | 7
Number of Seizures | 9 (2)
Statistical Analysis 1: Comparison: Thalidomide; Power=0.02; Test type: Non-Inferiority or Equivalence — p less than or equal to 0.05, repeated measures ANOVA; p < 0.02, ANOVA — p-value is non-adjusted for multiple comparisons; Was adjusted the degrees of freedom for the averaged test of significance; Mean Difference (Final Values) = 0.02 — The frequency of seizures at the beginning of the study and after treatment with thalidomide was contrasted in the same group patients

ADVERSE EVENTS:
Time Frame: 1 year
Description: During the trial we observed two serious adverse events, one of them presented exacerbation of seizures, another patient showed sedation, at 3 and 7 months respectively to the beginning of treatment.
  Other adverse events consisted in sensory neuropathy in 2 out of 7 patients tested with nerve conduction studies.
Arm/Group | Thalidomide
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 1/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thalidomide (N=7)
sedation (Nervous system disorders) | 1 (1)
seizures exacerbation (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thalidomide (N=7)
sensorial neuropathy (Nervous system disorders) | 1 (1) — Seven patients were in risk however two participant were affected with less adverse events consisted in sensory neuropathy tested with nerve conduction studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No